CLINICAL TRIAL: NCT03195127
Title: Development of a Rehabilitation Strengthening and Mobility Program for Ventilator Dependent Older Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Aging (NIA) (NIH); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Avelino Verceles, Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: HP-00047963; R03AG045100 (NIH)
Record Dates: First submitted 2017-06-16; First posted 2017-06-22 (Actual); Results first posted 2022-02-08 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Respiration, Artificial; Critical Illness; Chronic Disease; Exercise Therapy; Rehabilitation; Physical Therapy Modalities
Keywords: Physical Therapy Modalities; Rehabilitation; Exercise Therapy; Critical Illness; Respiration, Artificial; Chronic Disease
MeSH Terms: conditions — Respiratory Aspiration; Critical Illness; Chronic Disease

STUDY DESIGN:
Intervention Model Description: Up to 75 patients will be screened with a goal of enrolling 40 for participate in the intervention trial (20 in the multimodal treatment arm and 20 in a group receiving usual care).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- multimodal physical therapy (Experimental): Multimodal physical therapy sessions three times a week, for four weeks, lasting one hour. Consist of limb strengthening exercises, endurance training, and balance/coordination drills.
  Interventions: Other: multimodal physical therapy
- Usual care (No Intervention): Subjects will receive the standard therapy program provided by University Specialty Hospital therapy services. To compliment the physical therapy regimen, an optimized nutritional program will be administered according accepted guidelines.

INTERVENTIONS:
Other: multimodal physical therapy — Consist of limb strengthening exercises, endurance training, and balance/coordination drills. These exercises and training maneuvers may involve the use of handheld weights, nautilus weight equipment, elastic exercise bands, stationary exercise machines (recumbent exercise cycles, hand ergometer cycles), or treadmills. If the subject is fit enough, Tai Chi may be added to as a training method to help improve your balance and strength. In addition, the subject will be asked to wear an accelerometer on their wrist
  Arms: multimodal physical therapy

SUMMARY:
As the general population ages and technology advances, many who suffer from catastrophic critical illness (i.e. septic shock, respiratory failure, Acute Respiratory Disease Syndrome) survive only to find themselves severely physically debilitated and compromised from a pulmonary standpoint, requiring assistance from a mechanical ventilator in order to breath. Oftentimes, these patients require a long course of physical rehabilitation and ventilator support. These patients frequently remain ventilator dependent for greater than 3 weeks, and are thus referred to as requiring prolonged mechanical ventilation (PMV).

Older patients are at significantly higher risk for requiring PMV for reasons that are not entirely clear, but which may include physical deconditioning, impaired cardiopulmonary physiology, and cognitive or behavioral disturbances.

The purpose of this study is two fold: 1. to characterize the functional phenotype of ventilator dependent, and recently ventilated patients with respect to general strength, endurance, balance, and pulmonary functioning and body composition. 2. To pilot test a rehabilitation protocol that targets improving this populations disabilities through exercises focused on improving strength, endurance, balance, and pulmonary functioning.

DETAILED DESCRIPTION:
Screening will occur daily, at which time the subject's medical history and current condition will be reviewed. If they qualify informed consent will be obtained and the subject will undergo baseline tests of function and health.

The subject will be asked to perform simple tasks for baseline testing purposes. These include timed walking, lifting light weights or elastic exercise bands, assessment of handgrip strength, getting up out of a chair, breathing into a machine to test lung function, and answering questionnaires. The order of these tests may vary depending upon the subject's schedule and availability of equipment. It may be necessary to repeat one or more of the tests. Not all tests will be performed on everyone, depending upon one's strength, balance, coordination and endurance.

After the completion of the baseline tests subjects will be randomized into one of two groups. One group will receive a multimodal rehabilitation program (MRP) and usual care and the other will receive usual care physical therapy.

If the subject is randomized to the intervention group, he/she will receive special MRP sessions three times a week, for up to 8 weeks. Each session will last approximately one hour, and will consist of limb strengthening exercises, endurance training, and balance/coordination drills. These exercises and training maneuvers may involve the use of handheld weights, nautilus weight equipment, elastic exercise bands, stationary exercise machines (recumbent exercise cycles, hand ergometer cycles), or treadmills. All sessions will be supervised by a licensed physical therapist, physical trainer, or certified instructor, with a respiratory therapist present, if needed. Sessions will be conducted at the Pulmonary Rehabilitation Gymnasium at the University of Maryland, Midtown Campus (MTC) or in the subjects room at bedside.

If the subject is not randomized to the group receiving the MRP, they will receive the standard therapy program provided by MTC therapy services. To compliment the physical therapy regimen, an optimized nutritional program will be administered according accepted guidelines.

If the subject misses/does not complete a session the training period will be extended to insure completion of the required number of sessions. If the subject is not randomized to the group receiving the MRP, they will receive the standard therapy program provided by MTC therapy services.

After two weeks of additional training, or 6 MRP sessions, the subjects will be re-evaluated with repeat physical activity testing. The subject will be required to complete activities similar to what they performed during your baseline evaluation. Retesting will be conducted regardless of which training regimen the subject received (MRP vs. standard physical therapy). Subjects will then train for an additional 2 weeks followed by repeat testing.

The each subject's participation in the study will be completed 1) after eight weeks of physical therapy, 2) If the subject has been discharged from the Comprehensive Pulmonary Rehabilitation Unit, or MTC, 3) if the subject gets transferred from MTC.

All procedures will take place at MTC.

Exercises and maneuvers will include:

1. Limb strengthening exercises: various exercises will be conducted, both as assessment maneuvers, and as therapeutic purposes. These will include 1.lower extremity function (get up and go, sit to stand, isometric leg press/extension) 2. upper extremity function (modified military press, isometric triceps exercise, seated row, scapular depression).

   1. Isometric leg press/extension: Subjects will be asked to perform leg extension from a seated position against a pad attached to a machine that offers resistance. This resistance will be adjusted according to the force capability of each participant. The leg press maneuver will also be performed from a seated position.
   2. Modified military press: Subjects will be asked to perform this procedure from a seated position. A machine offering resistance will be gripped at shoulder level. The subject will be asked to extend their arms against the resistance to a straight position and then slowly lower the load until they are back in the starting position, with arms bent and hands at shoulder level.
   3. Isometric triceps exercise: From a seated position, a subject will be asked to hold a dumbell in one hand straight over their head with their back straight. the weight will be slowly lowered down behind the subjects neck in an arc with the elbow kept stationary. The subject will then press the bar upwards but re-extending their arm, thus completing the repetition upon full tricep extension.
   4. Tricep Press Exercise (as tolerated): Using an overhead pulley machine a subject will be asked to stand facing the machine holding the resistance bar in front of them at chest level with arms in a flexed position, palms facing away from them. The subject will then extend their arms in a downward motion, keeping the elbow stationary, until their arms are fully extended at the subjects side with palms facing backwards.
   5. Chest press: (Using dumbells or press machine as tolerated) The subject will lie on a bench or floor with a dumbbell in each hand, knees bent and your feet flat on the surface. The dumbells will be positioned shoulder width (in the laying position, directly above the shoulders) with arms and wrists straight and palms facing towards the subjects feet. To start a the exercise, the subject will lower the dumbells (or weight machine) towards their chest until the upper arms are at about a 45 degree angle to the body. The weights should lowered to a level approximately in line with the subjects chest. To complete the repetition, the subject is required to straighten their arms, concentrating on using their chest muscles until their arms are straight. The palms should face away from the patient, (or towards the patients feet) throughout the entire motion.
   6. Seated row: From a seated position, with their back and legs straight, the subject will be required to grasp the handle of the seated row pulley system with arms straight. Maintaining straight back and legs, the subject will pull the handle towards them, at waist level. The subject should concentrate on using their back muscles, rather than just their arms. Once the handle is pulled to the patients waist, the subject will slowly allow the handle to return to the starting position to complete the repetition.
   7. Scapular depression: (as tolerated) From a seated position keeping their back straight with arms and hands to each side, the subject will be asked to clasp the seat of the chair and lift their bottom from the seat by straightening your elbows and pushing the shoulders down. to complete the repetition, the subject will be lower him or herself slowly back to the seated starting position.

   The one repetition maximum (1 RM) will be measured on the same exercise equipment used for strengthening exercises at baseline and after the ST program. The 1 RM test is defined as the maximal resistance that can be moved through the full range of motion with proper form one time. The 1 RM maneuver will be performed for each limb strengthening exercise, and will be conducted and supervised by trained and licensed physical therapists. Ratings of perceived effort and discomfort will be recorded periodically throughout the test. The test will be immediately terminated if a high discomfort rating is reached during the test, which is unrelated to normal exertion-induced muscle fatigue.

   One-on-one supervision by qualified physical therapists will be used for all training sessions. These therapists will be able to demonstrate the proper technique and form for all exercise maneuvers. These exercises have been successfully performed in protocols completed by over 300 older men and women over the past several years, and are well-tolerated by participants. The investigators anticipate that all subjects will not be able to tolerate all tests, thus the testing regimen will be tailored to each subjects tolerance.
2. General strength (handgrip): The subject will be asked to perform this maneuver from a seated position with their upper arm and forearm at a 90 degree angle. Handgrip strength will be assess and recorded as the best of three attempts as measured on a dynamometer.
3. Maneuvers to assess pulmonary function, which include maximal expiratory pressure and maximal inspiratory pressure. All pulmonary function maneuvers are performed routinely at the USH pulmonary function laboratory by a trained respiratory therapist.

   1. Maximal Inspiratory Pressure (MIP) and Maximal Expiratory Pressure (MEP) are measurements aid in the evaluating for respiratory muscle weakness. MIP is the pressure generated during maximal inspiratory effort measured at the mouth. It is usually measured from residual volume (RV) (end of expiration). Inspiratory muscle strength is also inversely related to lung volume. Performing the maneuver requires the subject to exhale to RV. With tight seal at mouth and nose, inspire (using diaphragm) forcefully and sustain for 1-2 seconds.
   2. MEP is pressure generated during maximal expiratory effort measured at the mouth. It is measured at total lung capacity (TLC), (full breath). Expiratory muscle strength is directly related to lung volume. Performing the maneuver requires the subject to inhale to TLC. With tight seal at mouth and nose, expire (using diaphragm) forcefully and sustain for 1-2 seconds.
4. Six minute walk (Aerobic function): The subject will be asked to walk at their own pace on a 30 meter course outlined in a corridor at USH. Their total distance walked after six minutes will be recorded. During this test the patient will be continuously monitored using pulse oximetry, heart rate monitoring and subjective visual scales of dyspnea (borg index).
5. Balance and Gait: The Short Physical Performance Battery (SPPB) is a series of simple tests requiring the subject to perform repeated standing and sitting from a chair, stand in place with feet placed close to one another forming a narrow base, and to walk 4 meters. The SPPB has been well validated as a reproducible assessment of balance, gait speed and lower extremity strength and endurance, and has been used by the investigators in several studies without complication.
6. Skinfolds / Circumference measures: a tape measure will be used to measure the distance around one or more locations on the subjects body (for example: upper arm, thigh, waist, hips, chest). In addition, a skinfold caliper (measures skin thickness) will be used to assess body fat by gently pinching the skin at the same locations on the subjects body.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 or greater
* Received prolonged mechanical ventilation for >= 14 days during their last acute hospitalization
* Has received mechanical ventilation within the past 14 days for at least 6 hours in a 24 hour period
* Tracheostomy in place
* Subject is able to follow commands, and can give written or witnessed verbal consent in English
* Subject is eligible for physical rehabilitation
* All four limbs intact and mobile

Exclusion Criteria:

* Acute superimposed cardiopulmonary disease (ie.pulmonary edema, Stage IV congestive heart failure, COPD exacerbation, asthma attack, untreated infections, other)
* Severe functional impairment or physical impairment to rehabilitation
* Dementia, cognitive impairment (see attached description outlining cognitive impairment under additional documents)

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-06-28 (Actual); Primary Completion 2015-07-31 (Actual); Study Completion 2017-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Avelino C Verceles, MD,MS, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- U of Maryland, Baltimore, Professional Schools IRB, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Verceles AC, Wells CL, Sorkin JD, Terrin ML, Beans J, Jenkins T, Goldberg AP. A multimodal rehabilitation program for patients with ICU acquired weakness improves ventilator weaning and discharge home. J Crit Care. 2018 Oct;47:204-210. doi: 10.1016/j.jcrc.2018.07.006. Epub 2018 Jul 11. PMID 30025227

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Multimodal Physical Therapy | Usual Care
Started | 15 | 18
Completed | 15 | 17
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Multimodal Physical Therapy | Usual Care | Total
Number analyzed (Participants) | 15 | 17 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 12 | 22
  >=65 years | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (12.0) | 63.1 (11.4) | 60.3 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 8 | 10 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 9 | 9 | 18
  White | 6 | 8 | 14
Region of Enrollment [Number; unit: participants]
  United States | 15 | 17 | 32

OUTCOME MEASURES:

1. Primary Outcome: Functional Assessment: Handgrip
Description: Handgrip strength will be reported in kilograms
Time Frame: Upon completing of study, up to 56 days
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Multimodal Physical Therapy | Usual Care
Number analyzed (Participants) | 15 | 17
kg | 3.6 (5.4) | 1.3 (4.9)

2. Primary Outcome: Functional Assessment: Short Physical Performance Battery (SPPB)
Description: Short Physical Performance Battery will be reported as a score from 0 to 12 from with lower scores indicating a worse outcome
Time Frame: Upon Completion of study, up to 56 days
Population: Male and female survivors of critical illness all meeting criteria for ICU acquired weakness as defined by Stevens.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Multimodal Physical Therapy | Usual Care
Number analyzed (Participants) | 15 | 17
units on a scale | 3.6 (5.4) | 1.3 (4.9)

3. Primary Outcome: Functional Assessment: 4 Meter Gait Speed
Description: 4 meter gait speed will be reported in meters per second
Time Frame: Upon completion of study, up to 56 days
Measure: Mean (Standard Deviation); unit: m/s
Groups:
- Multimodal Physical Therapy: Exercise intervention group - 4 meter gait speed in meters per second.
- Usual Care: Control Group -4 meter gait speed in meters per second
Arm/Group | Multimodal Physical Therapy | Usual Care
Number analyzed (Participants) | 15 | 17
m/s | 0.13 (.16) | 0.07 (.20)

4. Primary Outcome: Functional Assessment: 6 Minute Walk Distance
Description: 6 minute walk distance will be reported in feet
Time Frame: Upon completion of study, up to 56 days
Measure: Mean (Standard Deviation); unit: feet
Groups:
- Multimodal Physical Therapy: Exercise intervention group distance walked in 6 minutes in meters
- Usual Care: Usual care group distance walked in 6 minutes in meters
Arm/Group | Multimodal Physical Therapy | Usual Care
Number analyzed (Participants) | 15 | 17
feet | 40.6 (65.1) | 19.9 (54.2)

5. Secondary Outcome: Percent of Patients Weaned From Mechanical Ventilation
Description: Proportion of patients weaned from mechanical ventilation expressed in percent of total in group
Time Frame: Upon completion of study, up to 56 days
Measure: Count of Participants; unit: Participants
Arm/Group | Multimodal Physical Therapy | Usual Care
Number analyzed (Participants) | 15 | 17
Participants | 13 | 7

6. Secondary Outcome: Percent of Patients Discharged Home
Description: Proportion of patients discharged home as a percentage of all patients in group
Time Frame: Upon completion of study, up to 56 days
Measure: Count of Participants; unit: Participants
Arm/Group | Multimodal Physical Therapy | Usual Care
Number analyzed (Participants) | 15 | 17
Participants | 8 | 2

ADVERSE EVENTS:
Arm/Group | Multimodal Physical Therapy | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/17
Other Adverse Events (participants affected / at risk) | 0/15 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes